CLINICAL TRIAL: NCT03022357
Title: Nigrosomal Iron Imaging in Parkinson's Disease
Acronym: N3iPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16048
Record Dates: First submitted 2017-01-04; First posted 2017-01-16 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2017-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Patient Outcome Assessment; ioflupane; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patient assessment — Clinical examination, Examination, Questionnaires
Radiation: DATScan — In small subgroup
Radiation: Orbital X-Ray — If foreign body in eye needs exclusion
Other: Magnetic Resonance Imaging (MRI) — MRI scanning of all subjects

SUMMARY:
Prospective observational study to compare sensitivity of 3T functional Magnetic Resonance Imaging (3T fMRI) at diagnosing Parkinson's Disease (PD) against the benchmark DaTScan diagnostic test and clinical diagnosis at follow up.

DETAILED DESCRIPTION:
Idiopathic Parkinson's is characterized by loss of midbrain dopaminergic neurons preferentially affecting the nigrosomes of the pars compacta of the substantia nigra (SNpc). At the time of clinical diagnosis, an estimated 50-70% of the neurons of the SNpc are lost. Non-invasive imaging of cell loss in the nigrosomes containing the SNpc dopaminergic neurons would be clinically desirable for accurate diagnosis in clinically uncertain cases of parkinsonism, especially in the early stages of Parkinson's. Investigators recently discovered that high resolution susceptibility weighted MRI at 7T and 3T demonstrates iron related signal loss of the NS1 in Parkinson's. These studies proved the feasibility and potential of in vivo nigrosome MRI as new diagnostic tool for Parkinson's. Further support of and confidence in our novel diagnostic concept comes from similar observations by other research groups.

Project goals To establish whether nigrosome MRI is an alternative to DatScanTM in the diagnosis of early Parkinson's in patients with diagnostic uncertainty.

To establish whether nigrosomal iron predicts the severity of Parkinson's. As a secondary aim the investigators will study if nigrosomal iron load as determined by susceptometry correlates to disease severity (MDS-UPDRS).

TRIAL / STUDY OBJECTIVES AND PURPOSE

PURPOSE

* To establish whether nigrosome MRI is an alternative to DatScan in the diagnosis of early Parkinson's
* To establish whether nigrosomal iron predicts the severity of Parkinson's.

PRIMARY OBJECTIVE Validation of NS1 MRI as a qualitative diagnostic marker in early Parkinson's

• To investigate whether the presence or absence of the swallow tail on nigrosome MRI at 3T is as accurate as DatScan and at least 80% sensitive and 80% specific to predict the final clinical diagnosis of Parkinson's vs. other movement disorder in patients with indeterminate or atypical parkinsonian features.

Hypothesis 1: That the swallow tail sign is an accurate marker of early Parkinson's

SECONDARY OBJECTIVES Biomarker discovery based on quantitative nigrosome iron markers in Parkinson's • To investigate whether diagnostic performance of nigrosome MRI can be further improved through quantitative assessment of nigrosomal iron and combination with neuromelanin metrics.

Hypothesis 2: That nigrosomal iron metrics further improve the detection of early Parkinson's

• To assess how well disease severity can be predicted by iron content in the nigrosome and by a combination of iron content and the size of the neuromelanin-rich nigra volume.

Hypothesis 3: That nigrosomal iron metrics are closely associated with severity of early Parkinson's

The investigators will be recruiting 145 patients with diagnostic uncertainty of Parkinson's Disease. These patients will undergo a MRI and DATscans and will be clinically examined. They will then be followed-up (clinical examination) in 12 months, identifying if they can be confirmed as having Parkinson's Disease, in order to compare the sensitivity and specificity of nigrosome1 detected by MRI with DATScan, potentially allowing a non-invasive and much less expensive means of diagnosing Parkinson's Disease.

ELIGIBILITY:
Inclusion criteria:

* Ability to give informed consent
* Age > 21 to < 90 years
* Clinical symptoms suspicious for a diagnosis of Parkinson's disease but clinical uncertainty with regards to a definite diagnosis:

  * Clinical symptoms not meeting all of the required UK brain bank diagnostic criteria for the diagnosis of PD
  * Clinical features not typically associated with PD and therefore raising the possibility of a different type disorder/movement disorder
* Referred for a DatScan as part of the NHS clinical diagnostic workup to investigate a suspicion for a parkinsonian movement disorder type disease or referred for a research DatScan as part of this study for the diagnostic workup to investigate a suspicion for a parkinsonian movement disorder type disease.

Exclusion criteria:

* Participants with any known contraindication to MRI such as:

  * Intracranial aneurysm clips
  * Cardiac pacemakers and defibrillators
  * Cochlear implants.
  * MR-incompatible metal implant or tattoo
  * Patients with a significant head tremor
  * Claustrophobia
  * Pregnant women
  * Participants that are felt to be unfit for the MRI scan according to the judgement of medically qualified personnel, either on the research team, or the patient's clinical team. (eg. due to back pain, claustrophobia, acute sickness etc.) This includes patients with signs of impaired temperature regulation such as an extremely high fever.
* (only for those planned for research DatScan) Participants in which a DatScan nuclear medical study can't be performed due to

  * Severe allergy to iodide compounds
  * Thyroid gland dysfunction

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potential participants need to have to capacity to give consent prior to study enrolment. Study participation is not possible if the participant is unable to give consent or does not have the capacity to consent.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of "swallow tail" on nigrosome MRI at 3T | 12 months
  Does absence of "swallow tail" on nigrosome MRI at 3T correlate with final diagnosis of Parkinson's Disease 12 months after initial presentation of clinically uncertain diagnosis? Is this correlation as accurate as that of DatScan? Is nigrosome MRI at 3T at least 80% sensitive and 80% specific to predict the final clinical diagnosis of Parkinson's disease vs. other movement disorders in patients with indeterminate or atypical parkinsonian features? Is the "swallow tail" and accurate marker of early Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee Auer (Principal Investigator), Principal Investigator — University of Nottingham; Stefan Schwarz (Co-Principal Investigator), Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Royal Derby Hospital, Derby, Derbyshire
  - Imperial College London, London
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarz ST, Afzal M, Morgan PS, Bajaj N, Gowland PA, Auer DP. The 'swallow tail' appearance of the healthy nigrosome - a new accurate test of Parkinson's disease: a case-control and retrospective cross-sectional MRI study at 3T. PLoS One. 2014 Apr 7;9(4):e93814. doi: 10.1371/journal.pone.0093814. eCollection 2014. PMID 24710392
- [Background] Blazejewska AI, Schwarz ST, Pitiot A, Stephenson MC, Lowe J, Bajaj N, Bowtell RW, Auer DP, Gowland PA. Visualization of nigrosome 1 and its loss in PD: pathoanatomical correlation and in vivo 7 T MRI. Neurology. 2013 Aug 6;81(6):534-40. doi: 10.1212/WNL.0b013e31829e6fd2. Epub 2013 Jul 10. PMID 23843466
- [Background] Cosottini M, Frosini D, Pesaresi I, Donatelli G, Cecchi P, Costagli M, Biagi L, Ceravolo R, Bonuccelli U, Tosetti M. Comparison of 3T and 7T susceptibility-weighted angiography of the substantia nigra in diagnosing Parkinson disease. AJNR Am J Neuroradiol. 2015 Mar;36(3):461-6. doi: 10.3174/ajnr.A4158. Epub 2014 Nov 6. PMID 25376811
- [Background] Reiter E, Mueller C, Pinter B, Krismer F, Scherfler C, Esterhammer R, Kremser C, Schocke M, Wenning GK, Poewe W, Seppi K. Dorsolateral nigral hyperintensity on 3.0T susceptibility-weighted imaging in neurodegenerative Parkinsonism. Mov Disord. 2015 Jul;30(8):1068-76. doi: 10.1002/mds.26171. Epub 2015 Mar 15. PMID 25773707
- [Background] Schuff N. Potential role of high-field MRI for studies in Parkinson's disease. Mov Disord. 2009;24 Suppl 2:S684-90. doi: 10.1002/mds.22647. PMID 19877239
- [Background] Piccini P, Whone A. Functional brain imaging in the differential diagnosis of Parkinson's disease. Lancet Neurol. 2004 May;3(5):284-90. doi: 10.1016/S1474-4422(04)00736-7. PMID 15099543
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Hughes AJ, Daniel SE, Ben-Shlomo Y, Lees AJ. The accuracy of diagnosis of parkinsonian syndromes in a specialist movement disorder service. Brain. 2002 Apr;125(Pt 4):861-70. doi: 10.1093/brain/awf080. PMID 11912118
- [Background] Rajput AH, Rozdilsky B, Rajput A. Accuracy of clinical diagnosis in parkinsonism--a prospective study. Can J Neurol Sci. 1991 Aug;18(3):275-8. doi: 10.1017/s0317167100031814. PMID 1913360
- [Background] Pirker W, Asenbaum S, Bencsits G, Prayer D, Gerschlager W, Deecke L, Brucke T. [123I]beta-CIT SPECT in multiple system atrophy, progressive supranuclear palsy, and corticobasal degeneration. Mov Disord. 2000 Nov;15(6):1158-67. doi: 10.1002/1531-8257(200011)15:63.0.co;2-0. PMID 11104200
- [Background] Fearnley JM, Lees AJ. Ageing and Parkinson's disease: substantia nigra regional selectivity. Brain. 1991 Oct;114 ( Pt 5):2283-301. doi: 10.1093/brain/114.5.2283. PMID 1933245
- [Background] Cosottini M, Frosini D, Pesaresi I, Costagli M, Biagi L, Ceravolo R, Bonuccelli U, Tosetti M. MR imaging of the substantia nigra at 7 T enables diagnosis of Parkinson disease. Radiology. 2014 Jun;271(3):831-8. doi: 10.1148/radiol.14131448. Epub 2014 Feb 26. PMID 24601752
- [Background] Kwon DH, Kim JM, Oh SH, Jeong HJ, Park SY, Oh ES, Chi JG, Kim YB, Jeon BS, Cho ZH. Seven-Tesla magnetic resonance images of the substantia nigra in Parkinson disease. Ann Neurol. 2012 Feb;71(2):267-77. doi: 10.1002/ana.22592. PMID 22367998
- [Background] Damier P, Hirsch EC, Agid Y, Graybiel AM. The substantia nigra of the human brain. I. Nigrosomes and the nigral matrix, a compartmental organization based on calbindin D(28K) immunohistochemistry. Brain. 1999 Aug;122 ( Pt 8):1421-36. doi: 10.1093/brain/122.8.1421. PMID 10430829
- [Background] Damier P, Hirsch EC, Agid Y, Graybiel AM. The substantia nigra of the human brain. II. Patterns of loss of dopamine-containing neurons in Parkinson's disease. Brain. 1999 Aug;122 ( Pt 8):1437-48. doi: 10.1093/brain/122.8.1437. PMID 10430830
- [Background] Baudrexel S, Nurnberger L, Rub U, Seifried C, Klein JC, Deller T, Steinmetz H, Deichmann R, Hilker R. Quantitative mapping of T1 and T2* discloses nigral and brainstem pathology in early Parkinson's disease. Neuroimage. 2010 Jun;51(2):512-20. doi: 10.1016/j.neuroimage.2010.03.005. Epub 2010 Mar 6. PMID 20211271
- [Background] Wallis LI, Paley MN, Graham JM, Grunewald RA, Wignall EL, Joy HM, Griffiths PD. MRI assessment of basal ganglia iron deposition in Parkinson's disease. J Magn Reson Imaging. 2008 Nov;28(5):1061-7. doi: 10.1002/jmri.21563. PMID 18972346
- [Background] Zhang W, Sun SG, Jiang YH, Qiao X, Sun X, Wu Y. Determination of brain iron content in patients with Parkinson's disease using magnetic susceptibility imaging. Neurosci Bull. 2009 Dec;25(6):353-60. doi: 10.1007/s12264-009-0225-8. PMID 19927171
- [Background] Beam CA. Strategies for improving power in diagnostic radiology research. AJR Am J Roentgenol. 1992 Sep;159(3):631-7. doi: 10.2214/ajr.159.3.1503041.
- [Derived] Schwarz ST, Xing Y, Naidu S, Birchall J, Skelly R, Perkins A, Evans J, Sare G, Martin-Bastida A, Bajaj N, Gowland P, Piccini P, Auer DP. Protocol of a single group prospective observational study on the diagnostic value of 3T susceptibility weighted MRI of nigrosome-1 in patients with parkinsonian symptoms: the N3iPD study (nigrosomal iron imaging in Parkinson's disease). BMJ Open. 2017 Dec 14;7(12):e016904. doi: 10.1136/bmjopen-2017-016904. PMID 29247084
- See also: NICE Guideline (UK). Diagnosing Parkinson's disease. 2006 [cited 2015 Jul 31] — http://www.ncbi.nlm.nih.gov/books/NBK48502/